CLINICAL TRIAL: NCT06222372
Title: Monitoring the Effect of Prophylactic Interventions in Contacts of Leprosy Patients Including Field-application of a Novel Immunodiagnostic Test in Bangladesh
Brief Title: Novel Interventions and Diagnostic Tests for Leprosy
Acronym: INDIGO#2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Annemieke Geluk (Other)
Collaborators: The Leprosy Mission Bangladesh (Other)
Responsible Party: Sponsor-Investigator, Annemieke Geluk, Prof. Dr. Annemieke Geluk, Leiden University Medical Center
Organization: Leiden University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: INDIGO#2
Record Dates: First submitted 2024-01-03; First posted 2024-01-24 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Leprosy
Keywords: leprosy, diagnostics, SDR, post exposure prophylaxis (PEP), biomarkers, UCP-LFA
MeSH Terms: conditions — Leprosy | interventions — Rifampin

STUDY DESIGN:
Intervention Model Description: Contacts of new MB leprosy patients with a bacterial index (BI) of 2 or more will be included. To determine the effect of SDR on M. leprae infection rate using UCP-LFA prospectively, SDR will be administered to 10 contacts of the new leprosy patients (n=100). M. leprae infection will be determined for each patient and contact by finger stick UCP-LFA for multiplex detection of anti-M. leprae antibodies and cytokines at time points 0 (intake), 2 weeks, 4 weeks, and 6 months after SDR (n=4,400). Contacts will include both household and neighbor contacts.
Who Masked: Participant
Masking Description: As an additional feature of this sub-study, we will test two SDR regimens. One regimen will be the until now standard SDR regimen of 600 mg rifampicin for adults weighing 35 kg and over, 450 mg for adults weighing less than 35 kg and for children older than 9 years, and 300 mg for children aged 5 to 9 years. The other regimen will be double this dose (1200 mg rifampicin for adults weighing 35 kg and over, 900 mg for adults weighing less than 35 kg and for children older than 9 years, and 600 mg for children aged 5 to 9 years). The patients and their contact group will be equally allocated through randomization to one of the two SDR regimen groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single dose rifampin (SDR) (Experimental): To household contacts of newly diagnosed leprosy patients SDR is provided as follows: 600 mg rifampicin for adults weighing 35 kg and over, 450 mg for adults weighing less than 35 kg and for children older than 9 years, and 300 mg for children aged 5 to 9 years.
  Interventions: Drug: Rifampin
- Single double dose rifampin (SDDR) (Experimental): To household contacts of newly diagnosed leprosy patients SDDR is provided as follows: 1200 mg rifampicin for adults weighing 35 kg and over, 900 mg for adults weighing less than 35 kg and for children older than 9 years, and 600 mg for children aged 5 to 9 years.
  Interventions: Drug: Rifampin

INTERVENTIONS:
Drug: Rifampin — antibiotic

SUMMARY:
Contact with Mycobacterium leprae (M. leprae) infected individuals is a risk factor for development of leprosy. Thus, detection of asymtomatically M. leprae infected individuals, allowing informed decision making on who needs treatment at a preclinical stage, is vital to interrupt transmission and can help prevent leprosy. In a previous field trial the BCG vaccine was applied alone and combined with a single dose of rifampin (SDR) as prophylactic interventions in contacts of leprosy patients in Bangladesh. Concurrently, blood-derived host immune-profiles specific for M. leprae infection or leprosy disease were assessed in the same population by merging detection of innate, adaptive cellular as well as humoral immunity. This has led to the identification of selected host-immune markers, currently applied in a low complexity lateral flow assay based on up-coverting particles (UCP-LFA), providing a convenient tool to assess M. leprae infection, allowing assessment of efficacy of prophylactic interventions in a point-of-care setting.

The proposed study aims to determine the effect of post-exposure prophylaxis by SDR on M. leprae infection rate using UCP-LFA before and after prophylaxis.

DETAILED DESCRIPTION:
A stable leprosy new case detection rate in many endemic countries indicates that the transmission of M. leprae is continuing unabated and that the current control strategy of case finding and provision of multi drug therapy (MDT) is not sufficient. Immunoprophylaxis by vaccination or post-exposure prophylaxis (PEP) with antibiotics provide effective strategies for the prevention of leprosy. Prophylactic treatment with single dose rifampicin (SDR) has shown to be a successful method to prevent leprosy in contacts of newly diagnosed leprosy patients (1). Currently, the Leprosy Post-Exposure Prophylaxis (LPEP) program generates evidence on the feasibility of integrating contact tracing and single-dose rifampicin (SDR) administration into routine leprosy control activities within the national leprosy control programmes of Brazil, Cambodia, India, Indonesia, Myanmar, Nepal, Sri Lanka and Tanzania [Steinmann P, et al]. Recently, the world health orginazation (WHO) has endorsed PEP for routine application in their new "Guidelines for the diagnosis, treatment and prevention of leprosy".

Genomic and transcriptomics analysis (e.g. population- and twin studies [5]), have determined that the host genetic background is an important risk factor for leprosy susceptibility. In addition, close contacts of leprosy patients have a higher risk of developing the disease (2, 3), which therefore represents the primary target group for interventions (4). To target individuals spreading leprosy bacilli for prophylactic treatment, M. leprae infection needs to be measurable objectively. Antibody levels correspond with bacterial load and risk of transmission. Also, individuals seropositive for anti-M. leprae phenolic glycolipid-I (PGL-I) antibodies, are at 5-8 fold higher risk of leprosy (5, 6). Moreover, in a leprosy endemic area in Bangladesh, we recently showed significant added value of cellular markers (cytokines, chemokines, acute phase proteins) to identify infection (7). Thus, for implementation in a PEP-approach, new tests that indicate who needs treatment should allow detection of both cellular-and humoral markers.

In previous studies applying UCP-LFA in 4 countries with variable leprosy endemicity (Bangladesh, Brazil, China and Ethiopia), we have shown that the combined assessment of serum levels of multiple biomarkers including anti-PGL-I Ab as well as cytokines, significantly improved the diagnostic potential for detection of M. leprae infected individuals. This demonstrates that UCP-LFAs for detection of multiple biomarkers can provide valuable tools for more accurate detection of M. leprae infection. Its low-complexity POC format and applicability for use of finger-stick blood allows large scale screening efforts in field settings. Moreover, the format of the UCP-LFA is being further developed in various other projects (focused on tuberculosis and leprosy diagnostic tests). This has recently resulted in a multi-biomarker test (MBT) format that allows simultaneous detection of up to 6 markers, which is currently further evaluated in the field for tuberculosis diagnostic purposes. Since the UCP-LFA format is flexible and can accommodate for detection of different markers, this latest development will also enable combined detection of humoral and cellular biomarkers which together represent a specific signature for M. leprae infection.

ELIGIBILITY:
Inclusion Criteria patients:

- newly diagnosed multibacillary leprosy patients (BI 1-6)

Inclusion Criteria contacts of MB leprosy patients:

* living in the same house (household members)
* living in a house on the same compound
* sharing the same kitchen
* direct neighbors (first neighbors)
* willing to participate
* provide informed consent

Exclusion Criteria patients:

* refusal of examination of their contacts
* suffering from the pure neural form of leprosy
* residing only temporarily in the study area
* PB leprosy patients

Exclusion Criteria contacts:

* diagnosed as leprosy patients during contact examination
* living less than 100 m away from a patient already included in the study
* first and second degree relatives of a patient already included in the study
* refusal informed consent
* pregnancy
* tuberculosis or leprosy treatment
* below 5 years of age
* known to suffer from liver disease or jaundice
* residing temporarily in the study area

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2020-03-04 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Changes of levels of host serum proteins in contacts after SDR | samples will be analysed 2 weeks, 4 weeks, and 6 months after SDR
  Using UCP-LFA levels of biomarkers will be quantified in fingerprick blood samples
Changes of levels of host serum proteins in contacts after SDDR | samples will be analysed 2 weeks, 4 weeks, and 6 months after SDDR
  Using UCP-LFA levels of biomarkers will be quantified in fingerprick blood samples

SECONDARY OUTCOMES:
Changes in bacterial load in contacts after SDR | samples will be analysed 2 weeks, 4 weeks, and 6 months after SDR
  determining M.leprae DNA in nasal swabs
Changes in bacterial load in contacts after SDDR | samples will be analysed 2 weeks, 4 weeks, and 6 months after SDDR
  determining M.leprae DNA in nasal swabs

CONTACTS AND LOCATIONS:
Overall Officials: Annemieke Geluk, PhD, Principal Investigator — Academisch Ziekenhuis Leiden (LUMC)
Locations (1):
- The Leprosy Mission International - Bangladesh, Nilphamari, Bangladesh

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-02-14): https://cdn.clinicaltrials.gov/large-docs/72/NCT06222372/ICF_000.pdf